CLINICAL TRIAL: NCT02041988
Title: Influence of Premedication With Oral Morphine Sulphate on Analgesic Consumption in Patient Undergoing Major Urological Surgery. Comparison Between Two Different Doses
Brief Title: Preemptive Analgesia With Morphine Sulphate in Major Urological Surgery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Francesco Cannata, Medical Doctor, University of Roma La Sapienza
Other Study IDs: 1846/08.04.10
Record Dates: First submitted 2013-07-01; First posted 2014-01-22 (Estimated); Last update posted 2014-01-22 (Estimated); Status verified 2014-01

CONDITIONS: Pain
Keywords: premedication; oral morphine; preemptive analgesia
MeSH Terms: conditions — Pain

STUDY DESIGN:
Observational Model: Case-Control
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 0,2 mg/kg oral morphine: Patients have been assigned to two groups of 20 individuals, they have been premedicated with oral morphine sulfate, 0,2 mg/kg group A, 0,4mg/kg group B.During surgery analgesic administration will be monitored
- 0,4 mg/ kg oral morphine: morphine and analgesic consumption throughout surgery will be monitored

SUMMARY:
In this study safety and efficacy of oral morphine sulphate is evaluated in order to reduce opioids administration during major urological surgery

DETAILED DESCRIPTION:
The administration of oral morphine sulfate could be useful to reduce the use of opioids in major urological surgery. This study aims to assess the safety and efficacy of two different oral morphine sulphate doses 0,2 mg/kg vs 0,4mg/kg in major urological surgery.

ELIGIBILITY:
Inclusion Criteria:

American Society of Anaesthesiologists physical status classification I/ II, age between 18 - 75, BMI 18 -30

Exclusion Criteria:

American Society of Anaesthesiologists physical status classification III/ IV, renal and hepatic insufficiency, postoperative nausea and vomiting after oral opioids administrations, neurological and psychiatric disorders.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients selected for major urological surgery
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2013-02; Primary Completion 2014-01 (Actual); Study Completion 2014-07 (Estimated)

PRIMARY OUTCOMES:
morphine sulphate consumption | six months

SECONDARY OUTCOMES:
vital signs | six months

OTHER OUTCOMES:
VAS score | six months
side effects | six months

CONTACTS AND LOCATIONS:
Overall Officials: Francesco MD Cannata, MD, Principal Investigator — Policlinico Umberto I
Locations (2):
- Italy (2):
  - Francesco Cannata, Rome, Rome
  - Policlinico Umberto I, Rome, Rome